CLINICAL TRIAL: NCT03453580
Title: Role of Multi Slice Computed Tomography Portography in Grading of Liver Cirrhosis
Brief Title: CT Portography in Grading of Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Hamza, principal investigator, Assiut University
Other Study IDs: MSCT GRADING
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-02

CONDITIONS: CT Portography Grading of Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: multislice computed tomography portography — imaging modality

SUMMARY:
Esophageal variceal bleeding and hepatic encephalopathy are serious complications of hepatic cirrhosis, and they may lead to high mortality rate and severely threaten life quality of the patients

DETAILED DESCRIPTION:
The occurrence and development of Esophageal variceal bleeding and hepatic encephalopathy are closely related with portal vein system diseases, such as collateral circulation of portal hypertension and portal vein thrombosis.

The prevention of Esophageal variceal bleeding and hepatic encephalopathy in hepatic cirrhosis has become a hot spot in clinical practice.

Three-dimensional reconstruction of images obtained by multi-slice spiral computed tomography portography (MSCTP) is clear, realistic, and accurate.

It can directly and quickly display all anatomical information of collateral portal vein system, and is recognized as a good method to display blood vessels

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and\or portal hypertension diagnosed by; laboratory or radiological parameters.

Exclusion Criteria:

* Patients with ligation, disconnection or shunting of esophageal varices. Patients with combined hepatic malignant tumor Patients with splenectomy. Patients with renal dysfunction or iodine allergy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-25 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Grading of liver cirrhosis | 15 min
  Grade I: i)level 4-5 by portal development will achieved in intrahepatic portal vein imaging; ii) collateral circulation mainly open at esophageal gastric fundus vein, or one branch of para-umbilical vein or esophageal peripheral vein was open; iii) hepatic artery-portal vein fistula or portal vein embolus was not formed.
  Grade II: i)level 3-4 by portal development will achieved in intrahepatic portal vein imaging; ii) in addition to opening of collateral circulation at esophageal gastric fundus vein, 2-3 branches of para-umbilical vein or esophageal peripheral vein open; iii) some hepatic artery-portal vein fistula or portal vein embolus not observed.
  Grade lll: level 2-3 by portal development are achieved in intrahepatic portal vein imaging; ii) esophageal gastric fundus vein, para-umbilical vein or esophageal peripheral vein all open, iii) hepatic artery-portal vein fistula or portal vein embolus is formed.
  Then we will do correlation with child -pugh score

SECONDARY OUTCOMES:
prediction of esophageal varices and hepatic encephalopathy | 20 min
  measuring diameters of main portal vein,left gastric, splenic, intra hepatic right and left portal vein.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Biecker E. Gastrointestinal Bleeding in Cirrhotic Patients with Portal Hypertension. ISRN Hepatol. 2013 Jul 22;2013:541836. doi: 10.1155/2013/541836. eCollection 2013. PMID 27335828
- [Result] Bajaj JS. Review article: potential mechanisms of action of rifaximin in the management of hepatic encephalopathy and other complications of cirrhosis. Aliment Pharmacol Ther. 2016 Jan;43 Suppl 1:11-26. doi: 10.1111/apt.13435. PMID 26618922
- [Result] Chu Q, Li Z, Zhang SM, Hu DY, Xiao M. Relationship between encephalopathy and portal vein-vena cava shunt: value of computed tomography during arterial portography. World J Gastroenterol. 2004 Jul 1;10(13):1939-42. doi: 10.3748/wjg.v10.i13.1939. PMID 15222041